CLINICAL TRIAL: NCT02971566
Title: Splanchnic Oxygenation and Perfusion Response to Enteral Feeds in Preterm Infants With Abnormal Antenatal Doppler: Pattern Assessment and Correlation With Feeding Intolerance
Brief Title: Splanchnic Oxygenation Response to Enteral Feeds in Preterm Infants With Abnormal Antenatal Doppler.
Acronym: AREDF-SO
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, University of Bologna (Italy), IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SO-2016-AREDF
Record Dates: First submitted 2016-11-19; First posted 2016-11-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Placental Insufficiency; NEC - Necrotizing Enterocolitis; Newborn, Premature; Feeding Disorder Neonatal
Keywords: feeding intolerance; preterm infants; near infrared spectroscopy; abnormal antenatal Doppler
MeSH Terms: conditions — Placental Insufficiency; Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gastrointestinal complications: Development of one ore more of the following gastrointestinal complications:
  * necrotizing enterocolitis (stage ≥2)
  * spontaneous intestinal perforation
  * feeding intolerance, defined as enteral feeding withholding ≥1 day because of suggestive clinical signs
- Controls: no evidence of gastrointestinal complications during the hospitalization

SUMMARY:
Antenatal absent or reversed end-diastolic flow (AREDF) velocity through the umbilical arteries places preterm infants at significant risk for developing gastrointestinal complications, such as feeding intolerance, necrotizing enterocolitis or spontaneous intestinal perforation. Due to the fear of the aforementioned conditions, the establishment of adequate enteral feeds is frequently hampered in this population. Previous postnatal Doppler studies have shown that AREDF preterm infants who later developed feeding intolerance have a decreased blood flow velocity in the superior mesenteric artery in response to the first enteral feed; to date, however, it is not known whether this hemodynamic impairment persists over time, or if it is associated with reduced splanchnic oxygenation and perfusion, monitored by Near-infrared spectroscopy (NIRS).

This observational prospective study aims:

* to assess the patterns of abdominal oxygenation and perfusion in response to enteral feeds in AREDF preterm infants at different phases of enteral feeding establishment;
* to evaluate a possible correlation with the development of gastrointestinal complications.

DETAILED DESCRIPTION:
Intrauterine growth restriction (IUGR) is a major cause of perinatal morbidity and mortality. Severe IUGR is often due to impaired placental circulation, with absent or reversed end-diastolic flow (AREDF) velocity through the umbilical arteries. Fetuses with AREDF adapt to chronic hypoxia by undergoing a blood flow redistribution, which favors cerebral perfusion at the expense of the mesenteric district. The resulting hypoxic-ischemic injury of the intestinal mucosa represents a major risk factor for the post-natal development of gastrointestinal complications, such as necrotizing enterocolitis (NEC), spontaneous intestinal perforation (SIP) and feeding intolerance (FI). Due to the fear of the aforementioned conditions, the establishment of adequate enteral feeding in AREDF preterm infants is often difficult; hence, the identification of infants at highest risk for GI complications could aid their delicate nutritional management.

Postnatal Doppler studies have shown a decreased blood flow velocity in the superior mesenteric artery in response to the first enteral feed in AREDF preterm infants who later developed feeding intolerance. A similar Doppler impairment and lower values of splanchnic oxygenation at feeding introduction have been described in non-IUGR preterm infants with later GI complications. To date, however, it is not known whether the impaired mesenteric blood flow observed after the first feed in high-risk AREDF infants persists over time, or if it correlates with reduced splanchnic oxygenation and perfusion.

This observational prospective study aims:

* to assess the patterns of abdominal oxygenation and perfusion in response to enteral feeds in AREDF preterm infants at different phases of enteral feeding establishment;
* to evaluate a possible correlation with the development of gastrointestinal complications.

Infants admitted to the Neonatal Intensive Care Unit (NICU) are consecutively enrolled in the study if fulfilling the following criteria: gestational age ≤34 weeks, stable clinical conditions, documented evidence of antenatal umbilical Doppler impairment.

Exclusion criteria are:

* Enteral feeding prior to the enrollment
* Major congenital abnormalities (including congenital heart diseases, gastroschisis, exomphalos)
* Hemodynamic instability, hypotension, patent ductus arteriosus, anemia, sepsis or other infections at time of NIRS monitoring

Written, informed consent to participate in the study is obtained from the parents/legal guardians of each infant before enrollment.

Enrolled infants undergo a continuous monitoring of splanchnic oxygenation (SrSO2) at enteral feeding introduction (15 ml/kg/die volumes administered within the first 48 hours of life) and full enteral feeding (FEF) achievement (enteral intake ≥150 ml/kg/die) from 30' before to 3 h after feed administration by means of INVOS 5100 oximeter (Somanetics Corporation, Troy, MI, USA).

A simultaneous monitoring of peripheral oxygen saturation (SpO2) is be performed in order to calculate splanchnic fractional oxygen extraction (SFOE) ratio ([SpO2-SrSO2]/SpO2). SrSO2 values recorded during hypoxic episodes (SpO2 <85%) are excluded from statistical analysis.

GI complications are defined as NEC stage ≥2, SIP and/or FI (enteral feeding withholding ≥1 day because of suggestive clinical signs). Enrolled infants are retrospectively divided into two groups: lack (group 1) vs. development (group 2) of GI complications.

Data are analyzed using IBM SPSS Statistic version 20.0.0 (IBM Corporation, IBM Corporation Armonk, New York, United States). Clinical characteristics in the study groups are compared by Mann-Whitney U test for continuous variables and chi-square test for categorical variables. Mann-Whitney U test is used to compare abdominal SrSO2 and FSOE patterns in response to feeds between groups 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* gestational age ≤34 weeks
* stable clinical conditions
* documented evidence of antenatal umbilical Doppler impairment
* written informed consent obtained from parents/guardians

Exclusion Criteria:

* Enteral feeding prior to the enrollment
* Major congenital abnormalities (including congenital heart diseases, gastroschisis, exomphalos)
* Hemodynamic instability, hypotension, patent ductus arteriosus, anemia, sepsis or other infections at time of NIRS monitoring

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 20 preterm infants admitted to the Neonatal Intensive Care Unit of Sant'Orsola-Malpighi University Hospital and fulfilling the inclusion criteria are going to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Increase/reduction of SrSO2 after enteral feeds | 3.5 hours
  Increase/reduction of SrSO2 values in response to enteral feeds in infants who have developed gastrointestinal complications during their hospitalization.

SECONDARY OUTCOMES:
Increase/reduction of FSOE after enteral feeds | 3.5 hours
  Increase/reduction of SrSO2 values in response to enteral feeds in infants who have developed gastrointestinal complications during their hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi T Corvaglia, Prof, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- Neonatal Intensive Care Unit of the S.Orsola-Malpighi Hospital, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kempley S, Gupta N, Linsell L, Dorling J, McCormick K, Mannix P, Juszczak E, Brocklehurst P, Leaf A; ADEPT Trial Collaborative Group. Feeding infants below 29 weeks' gestation with abnormal antenatal Doppler: analysis from a randomised trial. Arch Dis Child Fetal Neonatal Ed. 2014 Jan;99(1):F6-F11. doi: 10.1136/archdischild-2013-304393. Epub 2013 Aug 23. PMID 23973795
- [Background] Bora R, Mukhopadhyay K, Saxena AK, Jain V, Narang A. Prediction of feed intolerance and necrotizing enterocolitis in neonates with absent end diastolic flow in umbilical artery and the correlation of feed intolerance with postnatal superior mesenteric artery flow. J Matern Fetal Neonatal Med. 2009 Nov;22(11):1092-6. doi: 10.3109/14767050903029600. PMID 19900051
- [Background] Kempley ST, Gamsu HR, Vyas S, Nicolaides K. Effects of intrauterine growth retardation on postnatal visceral and cerebral blood flow velocity. Arch Dis Child. 1991 Oct;66(10 Spec No):1115-8. doi: 10.1136/adc.66.10_spec_no.1115. PMID 1750758
- [Derived] Martini S, Aceti A, Beghetti I, Faldella G, Corvaglia L. Feed-related Splanchnic Oxygenation in Preterm Infants With Abnormal Antenatal Doppler Developing Gut Complications. J Pediatr Gastroenterol Nutr. 2018 May;66(5):755-759. doi: 10.1097/MPG.0000000000001804. PMID 29112084